CLINICAL TRIAL: NCT06950645
Title: The Open-label Observation of Oral Hexavalent Reassorted Rotavirus Live Attenuated Vaccine (Vero Cell) in Healthy Adults and Children, as Well as the Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate Safety, Tolerability, and Immunogenicity in Healthy Infants
Brief Title: Clinical Trial on the Oral Hexavalent Reassortant Rotavirus Attenuated Live Vaccine (Vero Cells)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-RV-1001
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Phase I; sequential design; safety; tolerability; immunogenicity; Rotavirus gastroenteritis; vaccine

STUDY DESIGN:
Intervention Model Description: This study features a single-arm, open-label design for the adult and children groups, and a randomized, double-blind, placebo-controlled design for the infant group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking is only conducted for the infant group, while the adult and children group is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Adult (Experimental): The experimental vaccine will be administered in three doses, with a 28-day interval between each dose.
  Interventions: Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine
- Children (Experimental): The experimental vaccine will be administered in three doses, with a 28-day interval between each dose
  Interventions: Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine
- Infants low-dose 1 (Experimental): They will receive three low-dose experimental vaccine in a double-blind setting, with a 28-day interval between each dose.
  Interventions: Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine
- Infants low-dose 2 (Placebo Comparator): They will receive three doses of the placebo in a double-blind setting, with a 28-day interval between each dose
  Interventions: Biological: Placebo
- Infants high-dose 1 (Experimental): They will receive three high-dose experimental vaccine in a double-blind setting, with a 28-day interval between each dose
  Interventions: Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine
- Infants high-dose 2 (Placebo Comparator): They will receive three doses of the placebo in a double-blind setting,with a 28-day interval between each dose
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine — Oral hexavalent reassortant rotavirus attenuated live vaccine (high-dose) three doses administered orally
  Arms: Adult
Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine — Oral hexavalent reassortant rotavirus attenuated live vaccine (high-dose) three doses administered orally
  Arms: Children
Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine — Oral hexavalent reassortant rotavirus attenuated live vaccine (low-dose) three doses administered orally
  Arms: Infants low-dose 1
Biological: Placebo — Placebo of experimental vaccine for infants three doses administered orally
  Arms: Infants low-dose 2
Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine — Oral hexavalent reassortant rotavirus attenuated live vaccine (high-dose) three doses administered orally
  Arms: Infants high-dose 1
Biological: Placebo — Placebo of experimental vaccine for infants three doses administered orally
  Arms: Infants high-dose 2

SUMMARY:
The Phase I clinical trial of the oral hexavalent reassortant rotavirus attenuated live vaccine (Vero Cells) will be conducted in a population ranging from 6 weeks to 59 years of age.

The objective of this study is to evaluate the safety of investigational vaccine in healthy adults and children, as well as its safety tolerability, and immunogenicity in healthy infants.

The study will be an open-label observation in adults and children, and a randomized, double-blind, placebo-controlled clinical trial in infants.

DETAILED DESCRIPTION:
The Phase I clinical trial is an open-label observation involving healthy adults and children, as well as a randomized, double-blind, placebo-controlled study in healthy infants to evaluate the safety, tolerability, and immunogenicity of the investigaional vaccine. The investigational vaccine is available in both high-dose and low-dose formulations. The placebo is identical to the trial vaccine in all components except for the rotavirus.

This study will enroll 100 participants, consisting of 20 adults aged 18-59 years, 20 children aged 2-6 years, and 60 infants aged 6-12 weeks. Participants will be enrolled sequentially, starting with adults, followed by children, and then infants. Enrollment for the subsequent group will begin after a 14-day safety observation period and confirmation of acceptable safety in the preceding group. Adult and child participants will receive the investigational vaccine in an open-label manner. The infants will be enrolled into two cohorts of 30 participants each: a low-dose cohort and a high-dose cohort. Within each cohort, the infants will be randomly assigned to two groups at a ratio of 2:1 and will receive either the investigational vaccine or a placebo in a double-blind manner. The immunization schedule for both the vaccine and placebo consists of three doses administered at 28-day intervals.

Adverse events (AE) will be collected for all participants until 42 days after the last dose vaccination. Stool samples will be collected after each vaccination to detect vaccine strain shedding among infant participants. Serious adverse events (SAE) will be observed for 6 months from the last dose for adults and children or 12 months for infants. Blood samples from the infants will be collected at predetermined times to evaluate the immunogenicity of the investigational vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. The participant and/or their guardian is willing and able to comply with all study procedures, sign the informed consent form, and remain contactable throughout the study period.
2. Provide legal identification.
3. Male or female, aged 6 to 12 weeks, or 2 to 6 years, or 18 to 59 years, and in good health.
4. Fertile participants have no plans for pregnancy from the time of signing the informed consent form until 3 months after the last dose of the study vaccine and agree to use effective contraception, and have no plans for sperm or egg donation.

Exclusion Criteria:

1. Known allergy to the vaccine or its components, such as urticaria, dyspnea, angioedema, etc.
2. Current diarrhea or vomiting, or other gastrointestinal diseases, or having experienced gastroenteritis or any acute illness or acute exacerbation of chronic disease within the past 7 days, or those currently using antibiotics or antiviral therapy.
3. History of intussusception or chronic gastrointestinal disease, including gastrointestinal congenital anomalies that can easily cause intussusception (e.g., Meckel's diverticulum).
4. For infant and pediatric participants: congenital malformations or developmental disabilities, genetic defect diseases, severe malnutrition, or severe chronic diseases (such as Down syndrome, diabetes, sickle cell anemia, neurological disorders, Guillain-Barré syndrome); For adult participants: uncontrolled chronic diseases or severe disease history, including but not limited to cardiovascular diseases (such as drug-uncontrolled hypertension, i.e., systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg), hematologic diseases, hepatic and renal diseases, gastrointestinal diseases, respiratory diseases, malignant tumors, history of major organ transplantation, or any other disease or medical condition that the investigator believes may interfere with the trial results.
5. Presence of autoimmune diseases or immunodeficiency diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid disease, asplenia, functional asplenia, HIV infection).
6. Household members living with the participant are in an immunodeficient or immunosuppressed state or are currently/soon to be receiving immunosuppressive therapy, cytotoxic therapy, etc.
7. Presence of coagulation dysfunction (such as deficiency of coagulation factors, abnormal platelets).
8. Received >14 days of immunosuppressive therapy or other immunomodulatory therapy, cytotoxic therapy within the past 6 months (for adult and pediatric participants) or since birth (for infant participants), or planned to receive such treatment during the study period.
9. Chronic alcoholism [weekly alcohol consumption >14 drinking units (1 drinking unit = 14 grams of 100% alcohol = 360 mL beer, or 150 mL wine, or 45 mL distilled spirits/liquor)] or history of drug abuse (repeated, excessive use of narcotic drugs, psychotropic substances, volatile organic solvents, etc.) (for adult participants).
10. Suffering from/having suffered from severe neurological diseases (epilepsy, convulsions or seizures) or mental illness, or having a family history of the same.
11. Received immunoglobulin or other blood products within 6 months before receiving the trial vaccine (for adult and pediatric groups) or in the past (for infant group), or planned to receive such treatment during the study period.
12. Received other investigational drugs or vaccines within the past 30 days, or planned to receive such drugs or vaccines during the study period.
13. Received live attenuated vaccines or COVID-19 vaccines within the past 14 days, or subunit or inactivated vaccines and other process vaccines within the past 7 days.
14. Had axillary temperature ≥38.0℃ within the past 3 days.
15. On the day planned for vaccination with the trial vaccine, having a fever with axillary temperature >37.0℃.
16. Clinical laboratory tests showing laboratory abnormalities beyond the reference range that are clinically significant (for adult and pediatric groups):

    * Hematology test indicators: white blood cell count, hemoglobin, platelet count.
    * Biochemical blood test indicators: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), creatinine (CR), fasting blood glucose (Glu).
    * Urinalysis test indicators: urine protein (PRO).
17. Fertile women with positive urine pregnancy test or breastfeeding.
18. Currently or planning to participate in other vaccine or drug clinical trials.
19. Any other factors that the investigator deems unsuitable for participation in the clinical trial.

Additional Exclusion Criteria for Infants Aged 6 to 12 Weeks

1. Previously received rotavirus vaccine.
2. History of rotavirus infection.
3. Neonatal gestational age <37 weeks or ≥42 weeks.
4. Birth weight <2500g.
5. History of difficult labor, resuscitation from asphyxia, or neurological damage at birth.

Ages: 6 Weeks to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of the investigational vaccine | 0 day after the first dose till 42 days after the last dose
  Incidence of adverse events/reactions

SECONDARY OUTCOMES:
Evaluate the safety of the investigational vaccine | 0-14 days after each dose
  Incidence of adverse events/reactions
Evaluate the safety of the investigational vaccine | 0-30 minutes after each dose
  Incidence of adverse events/reactions
Evaluate the safety of the investigational vaccine in the healthy adults and children groups | day 3 after each dose
  Incidence of clinically significant abnormal laboratory parameters on day 3 after each dose in adult and children groups
Evaluate the safety of the investigational vaccine | Within 6 months after the last dose
  Incidence of serious adverse events (SAEs)
Evaluate the safety of the investigational vaccine in the healthy infant group | Within 12 months after the last dose in the infant group
  Incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs)
Evaluate the immunogenicity and immune persistence of the investigated vaccine in healthy infants. | 28 days after the full vaccination course
  Seroconversion rate of serum IgA antibodies against vaccine serotype rotavirus.
Evaluate the immunogenicity and immune persistence of the investigated vaccine in healthy infants. | 28 days after the full vaccination course
  Seropositivity rate of serum IgA antibodies against vaccine serotype rotavirus.
Evaluate the immunogenicity and immune persistence of the investigated vaccine in healthy infants. | 28 days after the full vaccination course
  Geometric mean concentration (GMC) of serum IgA antibodies against vaccine serotype rotavirus.
Evaluate the immunogenicity and immune persistence of the investigated vaccine in healthy infants. | 28 days after the full vaccination course
  Geometric mean increase (GMI) of serum IgA antibodies against vaccine serotype rotavirus.
Evaluate the immunogenicity and immune persistence of the investigated vaccine in healthy infants. | 6 months and 12 months after the full vaccination course
  Seropositivity rate of serum IgA antibodies against vaccine serotype rotavirus
Evaluate the immunogenicity and immune persistence of the investigated vaccine in healthy infants. | 6 months and 12 months after the full vaccination course
  Geometric mean concentration (GMC) of serum IgA antibodies against vaccine serotype rotavirus
Evaluate the fecal shedding of investigated vaccine strain in healthy infants after vaccination. | 0-14 days after each dose
  The shedding rate of the rotavirus vaccine strain in the stool.
Evaluate the fecal shedding of investigated vaccine strain in healthy infants after vaccination. | 0-14 days after each dose
  The shedding duration of the rotavirus vaccine strain in the stool.
Evaluate the reassortment and reversion of the rotavirus vaccine strain in stool samples of healthy infants after vaccination | 0-14 days after each dose,
  The incidence of reassortment and reversion of the rotavirus vaccine strain in stool samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided